CLINICAL TRIAL: NCT02008890
Title: A 52-week, Multicenter, Randomized, Double-blind, Placebo-controlled Study of Subcutaneous Secukinumab to Demonstrate Efficacy as Assessed by Palmoplantar Pustulosis Psoriasis Area and Severity Index (ppPASI) at 16 Weeks of Treatment, Compared to Placebo, and to Assess Long-term Safety, Tolerability, and Efficacy in Subjects With Moderate to Severe Chronic Palmoplantar Pustular Psoriasis - Amended With an Optional Extension Treatment Period of up to a Total of 148 Weeks
Brief Title: Palmoplantar Pustular Psoriasis Efficacy and Safety With Secukinumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A3301; 2013-003086-34 (EudraCT Number)
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Palmoplantar Pustular Psoriasis
Keywords: palmoplantar, pustular, psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Secukinumab 300mg (Experimental): Secukinumab 300mg once weekly at Weeks 1, 2 and 3, thereafter at 4-weekly intervals starting Week 4 until Week 48.
  In order to maintain the blinding beyond the primary endpoint, placebo was administered at Weeks 17, 18 and 19.
  For extension period: Secukinumab 300mg at 4-weekly intervals starting Week 52 up to Week 148.
  Interventions: Biological: Secukinumab 300mg; Biological: Placebo
- Secukinumab 150mg (Experimental): Secukinumab 150mg once weekly at Weeks 1, 2 and 3, thereafter at 4-weekly intervals starting Week 4 until Week 48.
  In order to maintain the blinding beyond the primary endpoint, placebo was administered at Weeks 17, 18 and 19.
  For extension period: Secukinumab 150mg at 4-weekly intervals starting Week 52 up to Week 148.
  Interventions: Biological: Secukinumab 150mg; Biological: Placebo
- Placebo (Placebo Comparator): Placebo once weekly at Weeks 1, 2 and 3, thereafter at 4-weekly intervals starting Week 4 until Week 12. Patients who achieved ppPASI 75 at Week 16 remained on placebo treatment Until week 48 and were not eligible to enter the extension. Patients who did not achieve ppPASI 75 at Week 16 were re-randomized to receive Secukinumab 150mg or Secukinumab 300mg from Week 16 onwards up to Week 148.
  Interventions: Biological: Secukinumab 300mg; Biological: Secukinumab 150mg; Biological: Placebo

INTERVENTIONS:
Biological: Secukinumab 300mg — Secukinumab was used as 150 mg pre-filled syringes (PFS) in a double-blinded fashion. Secukinumab 300 mg s.c. (two PFS injections of the 150 mg dose) self-administered
  Arms: Placebo; Secukinumab 300mg
Biological: Secukinumab 150mg — secukinumab 150 mg s.c. (one PFS injection of the 150 mg dose + one PFS injection of placebo) self-administered
  Arms: Placebo; Secukinumab 150mg
Biological: Placebo — secukinumab placebo s.c. (two PFS injections of placebo) self-administered

SUMMARY:
A one year study assessing the efficacy and safety of secukinumab compared with placebo in adult patients with moderate to severe palmoplantar pustular psoriasis - amended with an optional extension treatment period of up to a total of 148 weeks

ELIGIBILITY:
Inclusion Criteria:

* Palmoplantar pustular psoriasis for at least 6 months before Randomization
* Moderate to severe palmoplantar pustular psoriasis as defined at Baseline by:

  * ppPASI score of ≥ 12 and
  * DLQI ≥ 10
* Candidate for systemic therapy, defined as having palmoplantar pustular psoriasis inadequately controlled by:

  * Topical treatment, and/or
  * Phototherapy, and/or
  * Previous systemic therapy

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque psoriasis and pustular palmoplantar psoriasis (e.g., erythrodermic, guttate, or generalized pustular psoriasis)
* Drug-induced psoriasis (e.g., new onset or current exacerbation from beta-blockers, calcium channel inhibitors, or lithium) or history of proven contact dermatitis
* Patients not willing to limit UV light exposure (e.g. sunbathing and/or the use of tanning devices) during the course of the study
* Ongoing use of prohibited psoriasis treatments (e.g., topical or systemic corticosteroids, UV therapy). Washout periods detailed in the protocol have to be adhered to
* Previous exposure to any biologic drug directly targeting IL-17 or IL-17 Receptor (e.g., secukinumab, ixekizumab, or brodalumab)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment and for 16 weeks after stopping treatment
* Active ongoing inflammatory diseases other than psoriasis that might confound the evaluation of the benefit of secukinumab therapy
* Use of any other investigational drugs within 4 weeks of study drug initiation or within a period of 5 half-lives of the investigational treatment, whichever is longer

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2013-12-26 (Actual); Primary Completion 2014-11-24 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (64):
- Austria (4):
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- France (9):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Martigues
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse
- Germany (17):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanau
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mahlow
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Plauen
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Schwerin
- Italy (2):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
- Poland (4):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Zabrze
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Rostov on Don Region
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saratov
- Spain (5):
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Sweden (5):
  - Novartis Investigative Site, Gothenburg, Västra Götaland County
  - Novartis Investigative Site, Jönköping
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- United Kingdom (10):
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Dundee, Perthshire
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Portsmouth
  - Novartis Investigative Site, Wolverhampton
  - Novartis Investigative Site, York

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 337 patients were screened, and 237 of these patients completed the screening phase and were randomized to treatment.
Pre-assignment Details: At baseline patients were randomized at 61 study centers to one of the three treatment groups in a 1:1:1 ratio.
Groups:
- AIN457 150mg: Secukinumab 150mg at each dosing.
- AIN457 300mg: Secukinumab 300mg at each dosing.
- Placebo: Placebo at each dosing.
- Placebo - AIN457 150 mg: Placebo until Week 12. ppPASI 75 non-responder at Week 16. Secukinumab 150mg from Week 16 until the end of the study.
- Placebo - AIN457 300 mg: Placebo until Week 12. ppPASI 75 non-responder at Week 16. Secukinumab 300mg from Week 16 until the end of the study.
Period: Period 1
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Started | 80 | 79 | 78 | 0 | 0
Completed | 65 | 64 | 66 | 0 | 0
Not Completed | 15 | 15 | 12 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 7 | 5 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 6 | 8 | 6 | 0 | 0
Period: Period 2
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Started | 65 | 64 | 10 | 27 | 28
Completed | 38 | 49 | 9 | 13 | 20
Not Completed | 27 | 15 | 1 | 14 | 8
Not completed — Adverse Event | 12 | 7 | 0 | 5 | 5
Not completed — Withdrawal by Subject | 11 | 8 | 0 | 7 | 2
Not completed — Physician Decision | 4 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Period: Extension Period
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Started | 31 | 36 | 0 | 10 | 17
Completed | 26 | 31 | 0 | 6 | 13
Not Completed | 5 | 5 | 0 | 4 | 4
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 4 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- AIN457 150mg: Secukinumab 150mg at each dosing in period 1.
- AIN457 300mg: Secukinumab 300mg at each dosing in period 1.
- Placebo: Placebo at each dosing in period 1.
- Total: Total of all reporting groups
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo | Total
Number analyzed (Participants) | 80 | 79 | 78 | 237
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Randomized (Started)
  Years | 50.7 (13.68) | 50.6 (14.77) | 52.9 (11.33) | 51.4 (13.33)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Randomized (Started)
  Participants
    Female | 63 | 64 | 59 | 186
    Male | 17 | 15 | 19 | 51
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 1 | 0 | 1 | 2
  Caucasian | 78 | 78 | 76 | 232
  Missing | 1 | 0 | 1 | 2
  Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ppPASI 75 Response at Week 16 (Period 1)
Description: The primary endpoint was assessed by the palmoplantar pustulosis Psoriasis Area and Severity Index 75 (ppPASI 75). The percentage of subjects who achieved a 75% reduction in ppPASI score from Baseline to Week 16 was measured. The ppPASI is a modification of the PASI score and adjusted for palmoplantar pustular psoriasis by classifying and scoring erythema, scaling (desquamation) and pustules/vesicles. Both palms and both plants are scored from 0 to 4. The extent of involvement of each region of the body is scored from 0 to 6. The total ppPASI score can range from a lower level of 0, corresponding to no signs of psoriasis, up to a maximum of 72.
Time Frame: Baseline to Week 16
Population: Full Analysis Set (FAS = Started). A patient with a missing ppPASI assessment at Week 16 was considered as a responder if he/she has met the response criterion already at the time of drop-out. Otherwise he/she was considered as a non-responder.
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo
Number analyzed (Participants) | 80 | 79 | 78
percentage of participants | 17.5 | 26.6 | 14.1
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo; Test type: Superiority; p = 0.5722, Regression, Logistic; with factors treatment, country, body weight at baseline visit (> 90 kg or >= 90kg) and presence of plaque-type psoriasis; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.50 to 3.53]
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo; Test type: Superiority; p = 0.0411, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.04 to 6.60]

2. Secondary Outcome: ppPASI: Absolute Change From Baseline to Week 16
Description: A secondary endpoint was assessed by the palmoplantar pustulosis Psoriasis Area and Severity Index (ppPASI). The mean change of ppPASI score from Baseline to Week 16 was measured. The ppPASI is a modification of the PASI score and adjusted for palmoplantar pustular psoriasis by classifying and scoring erythema, scaling (desquamation) and pustules/vesicles. Both palms and both plants are scored from 0 to 4. The extent of involvement of each region is scored from 0 to 6. The total ppPASI score can range from a lower level of 0, corresponding to no signs of psoriasis, up to a maximum of 72.
Time Frame: Baseline to Week 16
Population: FAS - Including only Patients with ppPASI Scores at Baseline and Week 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo
Number analyzed (Participants) | 68 | 69 | 70
units on a scale
  Baseline | 21.79 (8.211) | 23.01 (10.787) | 23.10 (10.198)
  Change from Baseline to Week 16 | -6.99 (10.904) | -9.74 (12.130) | -6.73 (9.868)
Statistical Analysis 1: Comparison: AIN457 150mg vs Placebo; Test type: Superiority; p = 0.9431, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-4.59 to 3.47]
Statistical Analysis 2: Comparison: AIN457 300mg vs Placebo; Test type: Superiority; p = 0.1576, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.13, 95% CI 2-sided [-7.14 to 0.88]

3. Secondary Outcome: Percentage of Participants With ppPASI 75 Response Over Time (Period 1)
Description: A secondary endpoint was assessed as response rate of patients to treatment measured by the palmoplantar pustulosis Psoriasis Area and Severity Index 75 (ppPASI 75). The percentage of subjects who achieve a 75% reduction in ppPASI score from Baseline to each post-baseline visit is measured. The ppPASI is a modification of the PASI score and adjusted for palmoplantar pustular psoriasis by classifying and scoring erythema, scaling (desquamation) and pustules/vesicles. Both palms and both plants are scored from 0 to 4. The extent of involvement of each region of the body is scored from 0 to 6. The total ppPASI score can range from a lower level of 0, corresponding to no signs of psoriasis, up to a maximum of 72.
Time Frame: Baseline to Week 16
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo
Number analyzed (Participants) | 80 | 79 | 78
percentage of participants
  Week 1: number analyzed (Participants) | 79 | 79 | 75
  Week 1 | 0 | 1.3 | 1.3
  Week 2: number analyzed (Participants) | 79 | 78 | 77
  Week 2 | 1.3 | 1.3 | 0
  Week 3: number analyzed (Participants) | 78 | 74 | 71
  Week 3 | 2.6 | 5.4 | 0
  Week 4: number analyzed (Participants) | 77 | 77 | 74
  Week 4 | 6.5 | 9.1 | 1.4
  Week 8: number analyzed (Participants) | 77 | 75 | 73
  Week 8 | 13.0 | 13.3 | 9.6
  Week 12: number analyzed (Participants) | 75 | 71 | 69
  Week 12 | 14.7 | 23.9 | 10.1
  Week 16 | 17.5 | 26.6 | 14.1

4. Secondary Outcome: Percentage of Participants With ppPASI 75 Response Over Time (Period 2)
Description: as for outcome 3
Time Frame: Week 16 to Week 52
Population: FAS - Including only patients entering period 2
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 64 | 64 | 10 | 27 | 28
percentage of participants
  Week 16 | 18.8 | 31.3 | 90.0 | 0 | 0
  Week 20: number analyzed (Participants) | 64 | 64 | 10 | 26 | 28
  Week 20 | 20.3 | 31.3 | 80.0 | 7.7 | 17.9
  Week 24: number analyzed (Participants) | 63 | 64 | 10 | 26 | 26
  Week 24 | 30.2 | 37.5 | 80.0 | 19.2 | 38.5
  Week 32: number analyzed (Participants) | 55 | 58 | 10 | 20 | 25
  Week 32 | 36.4 | 48.3 | 80.0 | 25.0 | 44.0
  Week 40: number analyzed (Participants) | 45 | 55 | 10 | 16 | 24
  Week 40 | 44.4 | 56.4 | 70.0 | 37.5 | 50.0
  Week 48: number analyzed (Participants) | 42 | 50 | 10 | 15 | 19
  Week 48 | 52.4 | 58.0 | 60.0 | 40.0 | 47.4
  Week 52: number analyzed (Participants) | 38 | 51 | 9 | 14 | 20
  Week 52 | 57.9 | 58.8 | 66.7 | 50.0 | 60.0

5. Secondary Outcome: Percentage of Participants With ppPASI 75 Response Over Time (Extension Period)
Description: A secondary endpoint was assessed as response rate of patients to treatment measured by the palmoplantar pustulosis Psoriasis Area and Severity Index 75 (ppPASI 75). The percentage of subjects who achieved a 75% reduction in ppPASI score from Baseline to each post-baseline visit was measured. The ppPASI is a modification of the PASI score and adjusted for palmoplantar pustular psoriasis by classifying and scoring erythema, scaling (desquamation) and pustules/vesicles. Both palms and both plants are scored from 0 to 4. The extent of involvement of each region of the body is scored from 0 to 6. The total ppPASI score can range from a lower level of 0, corresponding to no signs of psoriasis, up to a maximum of 72.
Time Frame: Week 52 to Week 148
Population: FAS - Including only patients entering extension period (Placebo Week 16 responders not eligible)
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 31 | 36 | 10 | 17
percentage of participants
  Week 52 | 64.5 | 63.9 | 50.0 | 64.7
  Week 64: number analyzed (Participants) | 30 | 36 | 10 | 17
  Week 64 | 56.7 | 66.7 | 40.0 | 82.4
  Week 76: number analyzed (Participants) | 22 | 31 | 8 | 15
  Week 76 | 68.2 | 67.7 | 62.5 | 60.0
  Week 88: number analyzed (Participants) | 17 | 25 | 7 | 12
  Week 88 | 88.2 | 80.0 | 42.9 | 75.0
  Week 100: number analyzed (Participants) | 16 | 24 | 6 | 11
  Week 100 | 100.0 | 75.0 | 33.3 | 54.5
  Week 112: number analyzed (Participants) | 15 | 24 | 5 | 9
  Week 112 | 100.0 | 75.0 | 60.0 | 66.7
  Week 124: number analyzed (Participants) | 15 | 23 | 5 | 10
  Week 124 | 93.3 | 78.3 | 40.0 | 70.0
  Week 136: number analyzed (Participants) | 15 | 22 | 5 | 9
  Week 136 | 93.3 | 77.3 | 40.0 | 66.7
  Week 148: number analyzed (Participants) | 15 | 23 | 4 | 9
  Week 148 | 100.0 | 78.3 | 75.0 | 77.8

6. Secondary Outcome: Percentage of Participants With Most Frequent Adverse Events - Period 1 (Patient's Safety)
Description: Most frequent (at least 5% in any of the AIN457 groups) Adverse Events
Time Frame: Baseline to Week 16 (Period 1)
Population: Safety Set
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo
Number analyzed (Participants) | 80 | 79 | 78
percentage of participants
  Nasopharyngitis | 10.0 | 20.3 | 14.1
  Pustular psoriasis | 12.5 | 16.5 | 5.1
  Headache | 5.0 | 12.7 | 14.1
  Pruritus | 6.3 | 8.9 | 5.1
  Psoriasis | 6.3 | 5.1 | 3.8
  Urinary tract infection | 2.5 | 5.1 | 3.8
  Cough | 6.3 | 3.8 | 0
  Folliculitis | 3.8 | 5.1 | 1.3
  Nausea | 3.8 | 5.1 | 0
  Oral herpes | 5.0 | 1.3 | 0
  Rash pustular | 5.0 | 1.3 | 0

7. Secondary Outcome: Percentage of Participants With Most Frequent Adverse Events - Period 2 (Patient's Safety)
Description: Most frequent (at least 5% in any of the AIN457 groups) Adverse Events
Time Frame: Week 16 to Week 52 (Period 2)
Population: Safety Set - Including only patients entering period 2
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg | Placebo | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 64 | 64 | 10 | 27 | 28
percentage of participants
  Nasopharyngitis | 12.5 | 21.9 | 10.0 | 11.1 | 21.4
  Pustular psoriasis | 18.8 | 10.9 | 10.0 | 14.8 | 21.4
  Bronchitis | 4.7 | 9.4 | 0.0 | 3.7 | 10.7
  Headache | 4.7 | 6.3 | 0.0 | 3.7 | 7.1
  Eczema | 1.6 | 9.4 | 0.0 | 7.4 | 0.0
  Psoriasis | 3.1 | 4.7 | 20.0 | 7.4 | 0.0
  Pruritus | 3.1 | 4.7 | 10.0 | 0.0 | 7.1
  Folliculitis | 3.1 | 6.3 | 0.0 | 0.0 | 3.6
  Pain in extremity | 0.0 | 7.8 | 0.0 | 7.4 | 0.0
  Cough | 0.0 | 6.3 | 0.0 | 0.0 | 3.6
  Sinusitis | 0.0 | 1.6 | 10.0 | 7.4 | 3.6
  Skin infection | 1.6 | 3.1 | 0.0 | 7.4 | 0.0
  Urinary tract infection | 0.0 | 4.7 | 0.0 | 7.4 | 0.0
  Pruritus generalised | 1.6 | 1.6 | 0.0 | 7.4 | 0.0
  Rash | 0.0 | 6.3 | 0.0 | 0.0 | 0.0

8. Secondary Outcome: Percentage of Participants With Most Frequent Adverse Events - Extension Period (Patient's Safety)
Description: Most frequent (at least 5% in any of the AIN457 groups) Adverse Events
Time Frame: Week 52 to Week 148 (extension period)
Population: Safety Set - including only patients entering the extension period
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 150mg | AIN457 300mg
Number analyzed (Participants) | 41 | 53
percentage of participants
  Viral upper respiratory tract infection | 12.2 | 18.9
  Headache | 7.3 | 5.7
  Upper respiratory tract infection | 2.4 | 9.4
  Urinary tract infection | 9.8 | 3.8
  Diarrhoea | 4.9 | 5.7
  Tonsillitis | 2.4 | 5.7
  Ear infection | 7.3 | 0.0
  Oropharyngeal pain | 0.0 | 5.7

ADVERSE EVENTS:
Time Frame: Baseline to Week 148
Groups:
- Initial AIN457 150 mg: AEs for patients randomized to Secukinumab 150 mg at start of study.
- Initial AIN457 300 mg: AEs for patients randomized to Secukinumab 300 mg at start of study.
- Placebo: AEs for patients randomized to Placebo at start of study while treated with Placebo (AEs that occurred after re-randomization to Secukinumab are not counted in this group).
- AIN457 150 mg in Any Period: AEs for patients initially randomized to AIN457 150mg and placebo non-responder re-randomized to AIN457 150 mg at Week 16
- AIN457 300 mg in Any Period: AEs for patients initially randomized to AIN457 300mg and placebo non-responder re-randomized to AIN457 300 mg at Week 16
- Any AIN457: Any Secukinumab
Arm/Group | Initial AIN457 150 mg | Initial AIN457 300 mg | Placebo | AIN457 150 mg in Any Period | AIN457 300 mg in Any Period | Any AIN457
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/79 | 0/78 | 0/107 | 0/107 | 0/214
Serious Adverse Events (participants affected / at risk) | 9/80 | 13/79 | 5/78 | 11/107 | 17/107 | 28/214
Other Adverse Events (participants affected / at risk) | 73/80 | 73/79 | 53/78 | 92/107 | 94/107 | 186/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial AIN457 150 mg (N=80) | Initial AIN457 300 mg (N=79) | Placebo (N=78) | AIN457 150 mg in Any Period (N=107) | AIN457 300 mg in Any Period (N=107) | Any AIN457 (N=214)
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1 | 0 | 2 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 1 | 0 | 1 | 1 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Drug ineffective (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 0 | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Superinfection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 1 | 4 | 5
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial AIN457 150 mg (N=80) | Initial AIN457 300 mg (N=79) | Placebo (N=78) | AIN457 150 mg in Any Period (N=107) | AIN457 300 mg in Any Period (N=107) | Any AIN457 (N=214)
Bradycardia (Cardiac disorders) | 1 | 2 | 0 | 1 | 3 | 4
Tachycardia (Cardiac disorders) | 2 | 2 | 1 | 2 | 2 | 4
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 1 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 3 | 3 | 6
Aphthous ulcer (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 2 | 3
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 3 | 0 | 3
Dental caries (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 8 | 4 | 5 | 9 | 14
Nausea (Gastrointestinal disorders) | 3 | 6 | 0 | 4 | 7 | 11
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 2 | 4
Asthenia (General disorders) | 0 | 2 | 1 | 0 | 2 | 2
Chest pain (General disorders) | 2 | 1 | 1 | 2 | 1 | 3
Fatigue (General disorders) | 1 | 3 | 3 | 1 | 3 | 4
Feeling hot (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Injection site urticaria (General disorders) | 0 | 2 | 0 | 0 | 2 | 2
Pyrexia (General disorders) | 4 | 1 | 0 | 4 | 1 | 5
Drug hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 0 | 2 | 2
Bacterial vaginosis (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 2
Bronchitis (Infections and infestations) | 5 | 6 | 1 | 6 | 11 | 17
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 1 | 2 | 3
Conjunctivitis (Infections and infestations) | 4 | 3 | 0 | 4 | 4 | 8
Cystitis (Infections and infestations) | 3 | 1 | 1 | 4 | 2 | 6
Ear infection (Infections and infestations) | 1 | 0 | 0 | 4 | 0 | 4
Eczema impetiginous (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 2
Erysipelas (Infections and infestations) | 1 | 2 | 0 | 1 | 2 | 3
Folliculitis (Infections and infestations) | 5 | 8 | 1 | 5 | 9 | 14
Fungal skin infection (Infections and infestations) | 2 | 2 | 1 | 2 | 2 | 4
Furuncle (Infections and infestations) | 2 | 2 | 1 | 2 | 2 | 4
Gastroenteritis (Infections and infestations) | 2 | 3 | 0 | 2 | 3 | 5
Impetigo (Infections and infestations) | 0 | 2 | 0 | 0 | 2 | 2
Influenza (Infections and infestations) | 5 | 3 | 2 | 5 | 3 | 8
Laryngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 3 | 0 | 1 | 3 | 4
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 2 | 3
Oral candidiasis (Infections and infestations) | 0 | 5 | 2 | 0 | 5 | 5
Oral herpes (Infections and infestations) | 4 | 3 | 0 | 4 | 3 | 7
Otitis externa (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 2
Paronychia (Infections and infestations) | 2 | 1 | 0 | 2 | 1 | 3
Pharyngitis (Infections and infestations) | 3 | 1 | 0 | 4 | 1 | 5
Pharyngotonsillitis (Infections and infestations) | 1 | 2 | 0 | 1 | 3 | 4
Rash pustular (Infections and infestations) | 3 | 1 | 0 | 3 | 1 | 4
Sinusitis (Infections and infestations) | 1 | 3 | 1 | 3 | 4 | 7
Skin bacterial infection (Infections and infestations) | 3 | 3 | 1 | 3 | 4 | 7
Skin infection (Infections and infestations) | 1 | 2 | 1 | 3 | 2 | 5
Staphylococcal skin infection (Infections and infestations) | 3 | 1 | 0 | 3 | 1 | 4
Subcutaneous abscess (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 2
Tinea pedis (Infections and infestations) | 1 | 3 | 0 | 1 | 4 | 5
Tonsillitis (Infections and infestations) | 3 | 3 | 0 | 3 | 5 | 8
Tooth abscess (Infections and infestations) | 1 | 2 | 0 | 1 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 7 | 4 | 4 | 8 | 12
Urinary tract infection (Infections and infestations) | 5 | 5 | 3 | 7 | 6 | 13
Viral upper respiratory tract infection (Infections and infestations) | 17 | 31 | 12 | 20 | 40 | 60
Vulvovaginal candidiasis (Infections and infestations) | 1 | 3 | 1 | 1 | 3 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1 | 2 | 3
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1 | 2 | 2 | 4
Blood pressure increased (Investigations) | 1 | 2 | 0 | 1 | 2 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 2 | 0 | 2 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 3 | 0 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 1 | 3 | 4 | 1 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 5 | 6 | 4 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 4 | 5 | 8 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 4 | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 7 | 6 | 4 | 7 | 11
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2 | 0 | 2
Burning sensation (Nervous system disorders) | 0 | 1 | 2 | 0 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 2 | 2 | 4
Headache (Nervous system disorders) | 7 | 12 | 10 | 9 | 15 | 24
Migraine (Nervous system disorders) | 2 | 1 | 0 | 2 | 1 | 3
Sciatica (Nervous system disorders) | 2 | 3 | 2 | 2 | 4 | 6
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 3 | 3
Depression (Psychiatric disorders) | 3 | 1 | 2 | 3 | 1 | 4
Insomnia (Psychiatric disorders) | 1 | 2 | 2 | 1 | 2 | 3
Dysuria (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 2 | 2
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 3 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 0 | 5 | 9 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 2 | 6 | 8
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 1 | 4 | 5
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3 | 0 | 3
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 1 | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 0 | 2
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 3 | 7 | 3 | 5 | 7 | 12
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 2 | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 3 | 2 | 5
Lichen planus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 11 | 4 | 6 | 13 | 19
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 4 | 2 | 6
Psoriasis (Skin and subcutaneous tissue disorders) | 5 | 7 | 5 | 7 | 7 | 14
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 19 | 16 | 4 | 24 | 23 | 47
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 0 | 1 | 6 | 7
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 3 | 0 | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 1 | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 3 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 1 | 5 | 6
Hypertension (Vascular disorders) | 2 | 5 | 3 | 3 | 6 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.